CLINICAL TRIAL: NCT00791037
Title: Phase I/II Study of Adoptive T Cell Therapy Following In Vivo Priming With a HER-2/Neu (HER2) Intracellular Domain (ICD) Peptide-Based Vaccine in Patients With Advanced Stage HER2 Overexpressing Breast Cancer
Brief Title: Vaccine Therapy in Treating Patients With Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mary (Nora) Disis, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6658; NCI-2009-01591 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA129517 (NIH)
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-04

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Leukapheresis; Cyclophosphamide; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (vaccine therapy) (Experimental): Patients receive HER2/neu peptide vaccine admixed with sargramostim (GM-CSF) ID on days 1, 8, and 15. Beginning 2 weeks later, patients undergo leukapheresis to isolate and collect peripheral blood mononuclear cells for T-cell expansion.
  Patients receive cyclophosphamide IV once on day -1 and autologous ex vivo-expanded HER2-specific T cell IV over 30 minutes on day 1. Treatment repeats every 7-10 days for up to three immunizations. Patients receive a booster HER2/neu peptide vaccine 1 month after the final T-cell infusion, followed by 2 additional booster vaccines at 2-month intervals.
  Interventions: Biological: HER-2/neu peptide vaccine; Procedure: leukapheresis; Biological: ex vivo-expanded HER2-specific T cells; Drug: cyclophosphamide; Biological: sargramostim; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: HER-2/neu peptide vaccine — Given ID
  Other Names: HER-2
Procedure: leukapheresis — Undergo leukapheresis
Biological: ex vivo-expanded HER2-specific T cells — Given IV
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: sargramostim — Given ID
  Other Names: GM-CSF; Leukine; Prokine
Other: laboratory biomarker analysis — Correlative study

SUMMARY:
This phase I/II trial is studying the side effects of escalating doses of adoptive T cell therapy in treating patients with stage IV breast cancer. Vaccines are given to patient prior the expansion of a person's white blood cells may help the body build an effective immune response to kill tumor cells that overexpress human epidermal growth factor receptor 2 (HER2)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of infusing escalating doses of HER2 specific T cells into patients with advanced HER2+ breast cancer using ex vivo expanded autologous T cells.

SECONDARY OBJECTIVES:

I. To investigate to what extent HER2 specific T cell immunity can be boosted or generated in individuals after infusion of HER2 specific T cells.

II. To evaluate how long T cell immune augmentation persists in vivo after adoptive transfer of HER2 specific T cells and subsequent booster immunizations.

III. To determine the development of cluster of differentiation (CD)4+ and CD8+ epitope spreading after adoptive transfer of HER2 specific T cells.

TERTIARY OBJECTIVES:

I. To investigate the potential anti-tumor effects of HER2 specific T cells in patients with advanced HER2+ breast cancer.

II. To determine whether indium-labeled HER-2 specific T-cells traffic to sites of metastatic disease once adoptively transferred using SPECT or SPECT-CT imaging.

III. To assess whether adoptively transferred HER-2 specific T-cells induce acute inflammation at metastatic sites of disease by assessing the development of tumor inflammation after the second or third infusion of cells using PET-CT imaging.

OUTLINE: This is a phase I/II, dose-escalation study of ex vivo-expanded HER2-specific autologous T cells.

Patients receive HER2/neu peptide vaccine admixed with sargramostim (GM-CSF) intradermally (ID) on days 1, 8, and 15. Beginning 2 weeks later, patients undergo leukapheresis to isolate and collect peripheral blood mononuclear cells for T-cell expansion.

Patients receive cyclophosphamide intravenously (IV) once on day -1 and autologous ex vivo-expanded HER2-specific T cell IV over 30 minutes on day 1. Treatment repeats every 7-10 days for up to three treatments. Patients receive a booster HER2/neu peptide vaccine 1 month after the final T-cell infusion, followed by 2 additional booster vaccines at 2-month intervals.

While on the study, patients may continue their standard-of-care (non-research) treatment with trastuzumab and/or lapatinib IV weekly or every 3 weeks, except for 7 days before the cyclophosphamide dose, treatment 1 and treatment 2 and at least 7 days after receiving the second T cell vaccine. (Trastuzumab and lapatinib are not required or provided in this study).

Before the third T cell treatment of HER2 specific T-cells we will label a small sample of the patient's T-cells with indium-111. Prior to the final infusion of T-cells, patients will have FDG PET-CT performed. This scan will be repeated 48 hours after T-cell infusion. In addition, patients would then undergo SPECT or SPECT-CT imaging at 4, 24, 48, and 72 hours (+/- 3 hours) after labeled cells have been infused.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for the following year, and then twice a year thereafter. This consists of blood collection and contact with patients physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HER2+ Stage IV breast cancer that have been maximally treated and not achieved a complete remission
* Patients must have stable or slowly progressive disease state, measurable disease as:

  * Extraskeletal disease that can be accurately measured >= 10 mm by standard imaging techniques that can include but not limited to computed tomography (CT), positron emission tomography (PET), PET/CT, magnetic resonance imaging (MRI);
  * Skeletal or bone-only disease which is measurable by fludeoxyglucose (FDG) PET or PET/CT imaging will also be allowed
* Patients can be currently receiving trastuzumab and/or lapatinib and/or hormonal therapy and/or bisphosphonate therapy
* HER2 overexpression in the primary tumor or metastasis by immunohistochemistry (IHC) of 2+ or 3+, or documented gene amplification by fluorescence in situ hybridization (FISH) analysis; if overexpression is 2+ by IHC, then patients must have HER2 gene amplification documented by FISH
* Subjects must have a Performance Status Score (Southwest Oncology Group [SWOG]/Zubrod Scale) = 0, 1 or 2
* Patients must be off all immunosuppressive treatments such as chemotherapy or systemic steroid therapy a minimum of 14 days prior to initiation of study (i.e. first vaccination)
* Patients on trastuzumab and/or lapatinib must have a baseline left ventricular ejection fraction (LVEF) measured by multi gated acquisition scan (MUGA) or echocardiogram (ECHO) equal to or greater than the lower limit of normal for the facility within 90 days of eligibility determination
* Men and women of reproductive ability must agree to contraceptive use during the entire study period
* Patients must have an expected survival of 6 months
* White blood cell (WBC) >= 3000/mm^3
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Hemoglobin (Hgb) >= 10 mg/dl
* Platelets >= 75,000/mm^3
* Serum creatinine =< 2.0 mg/dl or creatinine clearance > 60 ml/min
* Total bilirubin =< 2.5 mg/dl
* Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) =< 3 times upper limit of normal (ULN)
* Patients must be >= 18 years old

Exclusion Criteria:

* Patients with any of the following cardiac conditions:

  * Symptomatic restrictive cardiomyopathy;
  * Unstable angina within 4 months prior to enrollment;
  * New York Heart Association functional class III-IV heart failure on active treatment
* Patients with any contraindication to receiving rhuGM-CSF based products
* Patients with any clinically significant autoimmune disease uncontrolled with treatment
* Patients with a history of brain metastases must have a stable head imaging study within 30 days of eligibility determination; specifically, patients with active brain metastases will not be eligible for study
* Patients who are simultaneously enrolled in any other treatment study
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-10; Primary Completion 2013-07 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Disis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
We will report study data but will not call out individual participants.

REFERENCES:
- [Derived] Stanton SE, Eary JF, Marzbani EA, Mankoff D, Salazar LG, Higgins D, Childs J, Reichow J, Dang Y, Disis ML. Concurrent SPECT/PET-CT imaging as a method for tracking adoptively transferred T-cells in vivo. J Immunother Cancer. 2016 May 17;4:27. doi: 10.1186/s40425-016-0131-3. eCollection 2016. PMID 27190628

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Vaccine Therapy+ex Vivo Expanded T Cells): Patients receive HER2/neu peptide vaccine admixed with sargramostim (GM-CSF) ID on days 1, 8, and 15. Beginning 2 weeks later, patients undergo leukapheresis to isolate and collect peripheral blood mononuclear cells for T-cell expansion.
  Patients receive cyclophosphamide IV once on day -1 and autologous ex vivo-expanded HER2-specific T cell IV over 30 minutes on day 1. Treatment repeats every 7-10 days for up to three immunizations. Patients receive a booster HER2/neu peptide vaccine 1 month after the final T-cell infusion, followed by 2 additional booster vaccines at 2-month intervals.
  HER-2/neu peptide vaccine: Given ID
  leukapheresis: Undergo leukapheresis
  ex vivo-expanded HER2-specific T cells: Given IV
  cyclophosphamide: Given IV
  sargramostim: Given ID
  laboratory biomarker analysis: Correlative study
Period: Overall Study
Arm/Group | Treatment (Vaccine Therapy+ex Vivo Expanded T Cells)
Started | 23
Primary Outcome | 19
Skeletal or Bone-only Disease by FDG-PET | 1
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Vaccine Therapy+ex Vivo T Cell Expansion): Patients receive HER2/neu peptide vaccine admixed with sargramostim (GM-CSF) ID on days 1, 8, and 15. Beginning 2 weeks later, patients undergo leukapheresis to isolate and collect peripheral blood mononuclear cells for T-cell expansion.
  Patients receive cyclophosphamide IV once on day -1 and autologous ex vivo-expanded HER2-specific T cell IV over 30 minutes on day 1. Treatment repeats every 7-10 days for up to three immunizations. Patients receive a booster HER2/neu peptide vaccine 1 month after the final T-cell infusion, followed by 2 additional booster vaccines at 2-month intervals.
  HER-2/neu peptide vaccine: Given ID
  leukapheresis: Undergo leukapheresis
  ex vivo-expanded HER2-specific T cells: Given IV
  cyclophosphamide: Given IV
  sargramostim: Given ID
  laboratory biomarker analysis: Correlative study
Arm/Group | Treatment (Vaccine Therapy+ex Vivo T Cell Expansion)
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Toxicity of Infusing HER2-specific T Cells as Assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0
Description: Patients are monitored for the development of end organ damage by assessing adverse events with serum chemistries, liver function studies, complete blood counts, urine analysis and physical exams. All adverse events for all systems are graded on a scale of 1-5 and attribution is assigned. There are DLT criteria. DLT is defined as any incidence of Grade 3 hematologic and non-hematologic toxicity (excluding: fever, hypoxia, and urticaria) Thus, if a subject develops a Grade 3 toxicity (excluding those listed in Table 4) will be considered excessive toxicity and no further dose escalations will occur.
Time Frame: Up to 4 months after first booster vaccine
Population: The infusion of escalating doses of HER2 specific T cells will be defined as safe if at least 75% of subjects are able to receive all 3 infusions without dose limiting toxicity (DLT)
Measure: Number; unit: participants
Groups:
- Treatment (Vaccine Therapy+ex Vivo-expanded T Cells): Patients receive HER2/neu peptide vaccine admixed with sargramostim (GM-CSF) ID on days 1, 8, and 15. Beginning 2 weeks later, patients undergo leukapheresis to isolate and collect peripheral blood mononuclear cells for T-cell expansion.
  Patients receive cyclophosphamide IV once on day -1 and autologous ex vivo-expanded HER2-specific T cell IV over 30 minutes on day 1. Treatment repeats every 7-10 days for up to three immunizations. Patients receive a booster HER2/neu peptide vaccine 1 month after the final T-cell infusion, followed by 2 additional booster vaccines at 2-month intervals.
  HER-2/neu peptide vaccine: Given ID
  leukapheresis: Undergo leukapheresis
  ex vivo-expanded HER2-specific T cells: Given IV
  cyclophosphamide: Given IV
  sargramostim: Given ID
  laboratory biomarker analysis: Correlative study
Arm/Group | Treatment (Vaccine Therapy+ex Vivo-expanded T Cells)
Number analyzed (Participants) | 19
participants | 0

2. Secondary Outcome: Proportion of Patients Whose T Cells Persist at a Level the Same or Greater as the Level After the Final T Cell Infusion and Subsequent Booster Immunizations as Assessed by IFN-gamma (IFN-g) ELISPOT
Time Frame: Up to 2 year following the last infusion
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Vaccine Therapy): Patients receive HER2/neu peptide vaccine admixed with sargramostim (GM-CSF) ID on days 1, 8, and 15. Beginning 2 weeks later, patients undergo leukapheresis to isolate and collect peripheral blood mononuclear cells for T-cell expansion.
  Patients receive cyclophosphamide IV once on day -1 and autologous ex vivo-expanded HER2-specific T cell IV over 30 minutes on day 1. Treatment repeats every 7-10 days for up to three immunizations. Patients receive a booster HER2/neu peptide vaccine 1 month after the final T-cell infusion, followed by 2 additional booster vaccines at 2-month intervals.
  HER-2/neu peptide vaccine: Given ID
  leukapheresis: Undergo leukapheresis
  ex vivo-expanded HER2-specific T cells: Given IV
  cyclophosphamide: Given IV
  sargramostim: Given ID
  laboratory biomarker analysis: Correlative study
Arm/Group | Treatment (Vaccine Therapy)
Number analyzed (Participants) | 19
Participants | 15

3. Secondary Outcome: Development of CD4+ and CD8+ Epitope Spreading
Description: As assessed by the development of immunity to epitopes within the HER2 protein to which the patient was not vaccinated as well as the development of immunity to other breast cancer related tumor antigens.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vaccine Therapy+ex Vivo Expanded T Cells)
Number analyzed (Participants) | 19
Participants | 12

4. Secondary Outcome: Response of Skeletal or Bone-only Disease by FDG-PET and According to European Organization for Research and Treatment for Cancer (EORTC)
Time Frame: Up to 2 years
Population: Due to getting regulatory approvals we could only enroll 1 patient in this part of the protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Vaccine Therapy+ex Vivo Expanded T Cells)
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 2 years and 6 months (Vaccine 1 through follow-up)*
Description: *The time between leukapheresis and first T cell infusion could vary due to patients being allowed to go back on treatment or scheduling conflicts.
Arm/Group | Treatment (Vaccine Therapy+ex Vivo Expanded T Cells)
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vaccine Therapy+ex Vivo Expanded T Cells) (N=23)
Unrelated Pulmonary Embolus (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Vaccine Therapy+ex Vivo Expanded T Cells) (N=23)
Abdominal pain (Gastrointestinal disorders) | 3 (4) — Pain
Alkaline phos increased (Investigations) | 2 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Alanine aminotransferase (Investigations) | 3 (3) — Increased
Anorexia (Metabolism and nutrition disorders) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6) — Arthralgia showed up various places: low back, R Hip, knee, joint
Aspartate aminotransferase increase (Investigations) | 8 (9) — Increase
Back pain (Musculoskeletal and connective tissue disorders) | 3 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (17)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 1 (2)
Non caridac chest pain (General disorders) | 4 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (9)
Diarrhea (Gastrointestinal disorders) | 7 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Lymphedema (Vascular disorders) | 6 (7)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 13 (17)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 (5)
Flu-like syndrome (General disorders) | 7 (10)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 1 (1)
Head/headache (Nervous system disorders) | 12 (25)
Anemia (Blood and lymphatic system disorders) | 13 (24)
Hot flashes/flushes (Vascular disorders) | 3 (3)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (4)
Hypertension (Vascular disorders) | 1 (1)
Urinary tract infections (Infections and infestations) | 3 (5)
Injection site reaction (General disorders) | 17 (52)
Insomnia (Psychiatric disorders) | 1 (1)
White blood cell decreased (Investigations) | 12 (17)
Lymphopenia (Investigations) | 13 (27) — lymphocyte count decrease
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (10)
Nausea (Gastrointestinal disorders) | 11 (17)
Neutrophil count decreased (Investigations) | 5 (9)
Upper respiratory infection (Infections and infestations) | 3 (4)
Lip infections (Infections and infestations) | 2 (3) — Herpes
Rigors/chills (General disorders) | 5 (10)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (14)
Platelets (Investigations) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6)
Proteinuria (Renal and urinary disorders) | 2 (2)
Pruritis/itching (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (5)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 12 (17)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (6)
Weight loss (Investigations) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Diaphoresis (Investigations) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2 (2)
Cardiac arrhythmia (Cardiac disorders) | 1 (1)
Creatinine (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Vericella zoster (General disorders) | 2 (2)
Axilla swelling/pain (Blood and lymphatic system disorders) | 1 (2)
Muscle pain (Musculoskeletal and connective tissue disorders) | 3 (3)
sensory neuropathy (Nervous system disorders) | 3 (3)
Body aches (General disorders) | 1 (1)
Pharyngitis/Rhinitis (Infections and infestations) | 1 (1)
Rash: Dermatitis associated with radiation (Injury, poisoning and procedural complications) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Left knee
Blood Disorders - Not clinically significant (Blood and lymphatic system disorders) | 10 (30)
Electrolyte Abnormalities - Not Clinically Significant (Metabolism and nutrition disorders) | 10 (20)
Non specific UA findings (Renal and urinary disorders) | 11 (68)

LIMITATIONS AND CAVEATS:
All Other Adverse Events are reported regardless of attribution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No